CLINICAL TRIAL: NCT07056283
Title: The Study of Urinary Biomarkers in Patients With Hypomagnesemia
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202500405
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Hypomagnesemia
Keywords: Hypomagnesemia; Magnesium

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypomagnesemia (serum Mg <1.7 mg/dL): The patients will be selected with a history of hypomagnesemia. The urine samples will be collected at various intervals depending on the most recent serum magnesium levels available during the study period. The patients may or may not be on medications known to alter serum magnesium levels.

SUMMARY:
In this pilot exploratory study, we aim to examine extracellular vesicles (EVs) as biomarkers in urine from up to 15 patients, with up to 10 samples per patient among the patients with a history of hypomagnesemia.

DETAILED DESCRIPTION:
Various medications (amiloride, SGLT2 inhibitors, calcineurin inhibitors) and medical conditions (type 2 diabetes mellitus, genetic factors) are associated with changes in blood magnesium levels, primarily by affecting magnesium transport in different regions of the kidney tubules. Over the past two decades, the discovery of extracellular vesicles (EVs) in urine has led to the emergence of a rapidly growing scientific field, offering an excellent non-invasive source for studying renal physiology. In this exploratory pilot study, we aim to enhance the mechanistic understanding of magnesium homeostasis by conducting noninvasive multi-omics (i.e., lipidomics, microRNAomics, and phospho-proteomics) research using urinary extracellular vesicles (uEVs) as biomarkers among patients with a history of hypomagnesemia. Fasting and post-magnesium-rich meal morning urine samples (6 am to 12 pm) will be collected at various intervals, depending on the most recent serum magnesium levels available during the study period. We will examine biomarkers capable of dissecting the mechanisms of hypomagnesemia.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years old)
* History of hypomagnesemia (serum Mg <1.7 mg/dL)

Exclusion Criteria:

* Current or recent use of loop, thiazide, or thiazide-like diuretics within the last 3 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient clinic patients at Shands Hospital, Gainesville, Florida, USA.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Changes in urinary markers pNKCC2/NKCC2, pNCC/NCC, pSPAK/SPAK, uEGF/Cr, TRPM6, Uromodulin | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Chintan Shah, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chacko KM, Nouri MZ, Schramm WC, Malik Z, Liu LP, Denslow ND, Alli AA. Tempol Alters Urinary Extracellular Vesicle Lipid Content and Release While Reducing Blood Pressure during the Development of Salt-Sensitive Hypertension. Biomolecules. 2021 Dec 1;11(12):1804. doi: 10.3390/biom11121804. PMID 34944449
- [Background] Lopez JP, Nouri MZ, Ebrahim A, Chacko KM, Schramm WC, Gholam MF, Ozrazgat-Baslanti T, Denslow ND, Alli AA. Lipid Profiles of Urinary Extracellular Vesicles Released during the Inactive and Active Phases of Aged Male Mice with Spontaneous Hypertension. Int J Mol Sci. 2022 Dec 6;23(23):15397. doi: 10.3390/ijms232315397. PMID 36499728
- [Background] Glover SC, Nouri MZ, Tuna KM, Mendoza Alvarez LB, Ryan LK, Shirley JF, Tang Y, Denslow ND, Alli AA. Lipidomic analysis of urinary exosomes from hereditary alpha-tryptasemia patients and healthy volunteers. FASEB Bioadv. 2019 Oct;1(10):624-638. doi: 10.1096/fba.2019-00030. Epub 2019 Aug 24. PMID 31803861
- [Background] Scindia YM, Gholam MF, Waleed A, Liu LP, Chacko KM, Desai D, Lopez JP, Malik Z, Schramm WC, Morales AG, Carson-Marino M, Alli AA. Metformin Alleviates Diabetes-Associated Hypertension by Attenuating the Renal Epithelial Sodium Channel. Biomedicines. 2023 Jan 21;11(2):305. doi: 10.3390/biomedicines11020305. PMID 36830842
- [Background] Schramm WC, Bala N, Arekar T, Malik Z, Chacko KM, Lewis RL, Denslow ND, Scindia Y, Alli AA. Enrichment of Bioactive Lipids in Urinary Extracellular Vesicles and Evidence of Apoptosis in Kidneys of Hypertensive Diabetic Cathepsin B Knockout Mice after Streptozotocin Treatment. Biomedicines. 2024 May 8;12(5):1038. doi: 10.3390/biomedicines12051038. PMID 38791000
- [Background] Aly R, Darwish S, Bala N, Ebrahim A, Shoemaker LR, McCray J, Garrett TJ, Alli AA. Functional and metabolomic analysis of urinary extracellular vesicles from juvenile mice with renal compensatory hypertrophy. Biochim Biophys Acta Mol Basis Dis. 2024 Jun;1870(5):167096. doi: 10.1016/j.bbadis.2024.167096. Epub 2024 Mar 16. PMID 38499276
- [Background] Pekkucuksen NT, Liu LP, Aly R, Shoemaker LR, Alli AA. Extracellular vesicles from focal segmental glomerulosclerosis pediatric patients induce STAT3 activation and mesangial cell proliferation. PLoS One. 2022 Nov 14;17(11):e0274598. doi: 10.1371/journal.pone.0274598. eCollection 2022. PMID 36374911